CLINICAL TRIAL: NCT06811168
Title: The Effect of Traditional Method and Kahoot! Gamification-Based Insulin Injection Training on Nursing Students' Knowledge, Skills, and Motivation Levels: A Randomized Controlled Study
Brief Title: The Effect of Traditional Method and Kahoot! Gamification-Based Insulin Injection Training on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, SEÇİL GÜLHAN GÜNER, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KaradenizTU-NURS-SGG-01
Record Dates: First submitted 2025-01-16; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Nurse's Role
Keywords: gamification; nurse; student; education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): the Kahoot! platform was introduced to the students and a mini trial test was conducted by the researchers who showed how to use it. Then, the Kahoot! (https://kahoot.it) application was downloaded to the students' mobile devices. The website was kept open throughout the study. One week after the theoretical training, each student logged into the system with a nickname and password they chose in the classroom environment. Students answered the Insulin Injection Knowledge Test-1 with Kahoot!. The answers given by the students and the score calculations were automatically recorded in the database.
  Interventions: Other: web based gamification
- No intervention (No Intervention): Insulin injection application was demonstrated to the students in the control group by the educator in a face-to-face training session supported by a PowerPoint presentation and video.

INTERVENTIONS:
Other: web based gamification — Kahoot gamificiation
  Arms: Experimental

SUMMARY:
This study was planned to examine the effects of insulin injection training using traditional methods and Kahoot! gamification on the knowledge, skills and motivation levels of participants.

DETAILED DESCRIPTION:
Technology, which we encounter in many areas of our lives, also affects the field of education in every aspect. Thanks to the use and development of technology, there are changes in the processes of accessing information and transferring information. In addition to current and technological changes in the process of transferring information, traditional and applied education are used in an integrated manner in nursing education. In the traditional education model used in nursing education, many problems are encountered such as many students receiving education together in crowded classes, insufficient use of demonstration methods, gaps between theory and practice in nursing education, and insufficient number of clinics. In this context, the problems experienced due to the education model used negatively affect the learning outcomes of the participants regarding nursing practices, and in this direction, it is envisaged that innovative education methods brought by technology will be used in nursing education. Insulin injection, which is one of the basic applications in nursing education, is frequently used in the treatment of diabetic patients as theoretical education and practice and is applied by nurses. Due to application errors in subcutaneous insulin injection, glycemic balance cannot be achieved in diabetic patients and may cause delays in the treatment process. Therefore, factors such as selecting the right application area for insulin injection, its correct application, and correct adjustment of insulin dose are very important in diabetes management. Insulin injection application and patient education on this subject are primarily the responsibility of nurses and all other health professionals. Within the scope of nursing education, all other applications such as insulin injection application are taught to participants theoretically, in laboratory and clinical environments, by researchers, through demonstration and laboratory practice, if possible. However, due to the high number of participants in nursing departments, insufficient number of researchers and most laboratory environments not having the facilities of real hospital environments, some information, skills and applications cannot be fully learned by the participants. In this context, it should be a priority in nursing education for the participants to perform the applications safely and to repeat them before going to the clinical environment, thus eliminating threats to patient safety. At the same time, an entertaining, educational and repetitive education environment should be created for the participant. Therefore, learning environments should be enriched by using information technologies in traditional learning methods and skill applications. Today, the web-based education approach is frequently used in the use of technology in nursing education. Web-based education is known as a student-centered approach that encourages lifelong learning through the use of information and communication technologies. The benefits of web-based education for participants include providing them with the responsibility of self-learning, making them aware of correct and incorrect information/applications, having participants do applications that they cannot do virtually, and providing them with the habit of lifelong learning. When the studies in the literature are examined, it is emphasized that the use of the web-based education approach in nursing education has positive effects on the cognitive and psychomotor levels of participants, academic success scores in courses, motivation and self-confidence levels. Kahoot!, one of the game-based learning platforms used in the web-based education process; is an online game tool where researchers can develop and share interactive exams, surveys, case studies, presentations and games in educational environments. In this platform, participants participate online via tablet, phone or computer and answer the prepared questions. With Kahoot!, participants are evaluated faster and more practically by educators thanks to the platform, their deficiencies/wrong answers are examined and they are guided to reach the correct answers. In addition, it has been seen that the use of this platform in the field of education increases the motivation of the participants and contributes positively to their learning performance and concentration. When the literature is examined, no study was found that evaluates the knowledge, skills and motivation of the participants in insulin injection education using traditional methods and game-based education approaches in nursing students, therefore this study is original. Especially in web-based education in nursing education, learning based on the game-based teaching approach allows both theoretical education and case analysis on the subject and is a method that is becoming widespread in the provinces. In the light of this information, it is thought that the use of Kahoot! gamification in addition to traditional education methods will contribute to the field of nursing education. In this context, this study was planned to examine the effects of insulin injection education given using traditional methods and Kahoot! gamification on the knowledge, skills and motivation levels of the participants. For this purpose, the hypotheses of the research are; H1: Insulin injection training provided with traditional methods has an effect on the knowledge level of the participants.

H2: Insulin injection training provided with traditional methods has no effect on the knowledge level of the participants.

H3: Insulin injection training provided with traditional methods has an effect on the skill level of the participants.

H4: Insulin injection training provided with traditional methods has no effect on the skill level of the participants.

H5: Insulin injection training provided with traditional methods has an effect on the motivation level of the participants.

H6: Insulin injection training provided with traditional methods has no effect on the motivation level of the participants.

H7: Kahoot! insulin injection training with gamification has an effect on the knowledge level of the participants.

H8: Kahoot! insulin injection training with gamification has no effect on the knowledge level of the participants.

H9: Kahoot! insulin injection training with gamification has an effect on the skill level of the participants.

H10: Kahoot! insulin injection training with gamification has no effect on the skill level of the participants.

H11: Kahoot! Insulin injection training with gamification has an effect on the motivation level of the participants.

H12: Kahoot! insulin injection training with gamification has no effect on the motivation level of the participants.

The universe of the study consists of 160 participants enrolled in the 2nd year Internal Medicine Nursing course of the Nursing Department of the Faculty of Health Sciences of Karadeniz Technical University. Power analysis was performed to determine the number of participants to be included in the study. The power of the test was calculated with the G*Power 3.1 program. As a similar study in the relevant literature, the effect size regarding the knowledge level difference was calculated as 0.789. In order to exceed the 95% value in determining the power of the study; 72 people and 36 groups need to be reached at a significance level of 5% and an effect size of 0.789 (df=70; t=1.667). Considering the high power of the test and the losses in the study, it was aimed to reach a total of 88 participants in 44 groups. Randomization will be performed in order to prevent bias in the people to be included in the study.

Inclusion criteria for the study:

* Those taking the Internal Medicine Nursing course for the first time,
* Those who own a computer or smartphone,
* Those who have uninterrupted internet access.

Inclusion criteria for the study:

* Those who have previously received insulin injection training,
* Those who have graduated from a health vocational high school,
* Those who are taking the Internal Medicine Nursing course for the second time due to failure, and
* Participants who are absent during the study will not be included in the study.

Data for the study will be collected using the "Participant Information Form", "Insulin Injection Success Test-1", "Insulin Injection Skill Control Test", "Motivation Scale for Teaching Materials" and "Insulin Injection Success Test-2".

ELIGIBILITY:
Inclusion Criteria:

* Taking the Internal Medicine Nursing course for the first time,
* Having a computer or smart phone,
* Having uninterrupted internet access.

Exclusion Criteria:

* Having received insulin injection training before,
* Having received training in a health-related department before,
* Taking the Internal Medicine Nursing course for the second time due to failure,
* Being absent at the time the research was conducted.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Knowledge | two weeks
  These data were collected with "Insulin Injection Knowledge Test-1 an Test-2". It was prepared to evaluate the knowledge level of students about insulin and insulin injection. The test consists of a total of 20 multiple choice questions covering theoretical knowledge about insulin and case analysis. The highest score that can be obtained from the entire test is 100, and the lowest score is 0. As the score increases, the level of knowledge increases.

SECONDARY OUTCOMES:
Skills | one weeks
  These data were collected with "Insulin Injection Skill Control Test". In order to examine students' psychomotor skills, the insulin injection skill checklist was prepared as 10 items. The application stages were scored as "0" if the skill was not present or was incorrect, or "10" if the skill was performed correctly. Therefore, the minimum score of the insulin injection skill checklist is "0", while the maximum score is "100".

OTHER OUTCOMES:
Motivation | two weeks
  These data were collected with "Motivation Scale for Teaching Materials". It is a measurement tool with 33 items, a five-point Likert type, and four sub-dimensions. The highest score that can be obtained from the entire scale is 165, and the lowest score is 33. The highest score that can be obtained from the attention dimension is 50, and the lowest score is 10. The highest score that can be obtained from the suitability dimension is 40, and the lowest score is 8. The highest score that can be obtained from the trust dimension is 45, and the lowest score is 9. The highest score that can be obtained from the satisfaction dimension is 30, and the lowest score is 6. An increase in the score obtained from the scale is interpreted as an increase in motivation towards the teaching material.

CONTACTS AND LOCATIONS:
Overall Officials: Seçil GÜLHAN GÜNER, PhD, Principal Investigator — Karadeniz Technical University
Locations (1):
- Seçil Gülhan Güner, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No